CLINICAL TRIAL: NCT06850961
Title: A Digital Health Intervention for Promoting Self-management in Patients With Chronic Obstructive Pulmonary Disease - a Feasibility Study
Brief Title: A Digital Health Intervention to Promote Self-management in Patients With Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Collaborators: Helse Forde (Other)
Responsible Party: Principal Investigator, Bente Frisk, Professor, Western Norway University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK2024/733856; REK2024/733856 (Other: Western Norway Regional Committees for Medical and Health Research Ethics)
Record Dates: First submitted 2024-12-02; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Self-management; Mobile Application; Feasibility Studies
Keywords: COPD; Digital health intervention; Feasibility; Self-management; Mobile Application
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The investigators will use the mobile app "Pust Deg Bedre" to explore the feasibility and experiences of providing PDB for patients with COPD,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital health intervention group (Experimental): Patients with COPD will use the mobile-app in self-management of treating dyspnea and mucus secretion.
  Interventions: Device: Digital health intervention by using a mobile application; Other: Feasibilty study and qualitative interview studies

INTERVENTIONS:
Device: Digital health intervention by using a mobile application — A digital health intervention for promoting self-management in patients with COPD by using a mobile application.
Other: Feasibilty study and qualitative interview studies — This study is a one group feasibility study including quantitative and qualitative study designs. The investigators will use focus groups and indiviual interviews, as well as Interpersonal Process Recall (IPR) interviews.

SUMMARY:
Dyspnea, cough, and chronic mucus hypersecretion are common symptoms in patients with Chronic Obstructive Pulmonary Disease (COPD), which increases risk of infections followed by exacerbations, often leading to hospitalization, disease progression and mortality. This patient group requires lifelong treatment in healthcare. A mobile application was developed to facilitate adherence to evidence-based guidelines for tailored breathing and airway clearance techniques to enhance self-management. The app is only in Norwegian and has a Norwegian name which is "Pust Deg Bedre" (PDB). The PDB app is fully developed and tested and can be downloaded for free. The app seems promising as a treatment tool, but has not yet been clinical evaluated. This project aims to 1) explore the feasibility of providing the app for patients with COPD, 2) explore the patients' with COPD experiences with the use of the PDB-app in treating dyspnea and mucus secretion, 3) explore the physiotherapists' experiences with the use of the PDB-app in treating dyspnea and mucus secretion, 4) explore the physiotherapists' experiences with implementing the PDB-app in treatment of patients with COPD, 5) explore the patients' experiences with the education in use of the PDB-app, and 6) At a 6-month follow up: explore the physiotherapists experiences with the usefulness and applicability of PBD-app, and to generally explore their experiences with participating in the project.

DETAILED DESCRIPTION:
This project is designed to explore aspects of acceptability and possible uncertainties associated with implementing the PDB-app as part of self-management in patients with COPD. Both quantitative and qualitative data will be collected and analysed.

50-60 patients with COPD and 15-30 physiotherapists in primary health care will be recruited.

A feasibility study will be conducted and evaluated after 8-week intervention and at 6-month follow-up, using a pre-post design.

Intervention: The physiotherapists will be responsible for providing the patients with training on the use of the PDB-app. Based on clinical assessment, the patients will receive a tailored treatment plan within the app. Patients are expected to engage with the tailored PDB-treatment for 8 weeks with follow-up after 6 months. If necessarily, adjustments to the treatment plan will be made throughout the intervention period. Follow-up of patients will occur digitally and physically.

A qualitative interview study will be conducted with semi-structured interviews after 8 weeks of intervention for a deeper understanding of the patients' and physiotherapists' experiences with the PDB-app. Separate focus groups will be conducted with the patients and the physiotherapists.

The investigators will also conduct video-recorded physiotherapy sessions at two time points during the intervention. The first one during the initial session, and then again between 3 to 6 weeks during the 8-week intervention. Subsequently, in-depth interviews, using Interpersonal Process Recall (IPR), will be conducted, with the researcher and physiotherapist, and with the researcher and patient. By using IPR interviews, video-assisted recall will help research participants access underlying experiences of their recent clinical interactions and put them into words. This means that the interaction between patient, physiotherapist and the PDB-app, experienced and recalled in the interview, relates to concrete events of the specific session.

Targeting physiotherapists, the investigators aim to do a long-term follow up 6 months after the intervention and explore their experiences with having participated in IPR interviews and as participants in the study in general. How and to what degree has the IPR interview sessions and the experiences from participating in this project impacted on their clinical practice, perception of role, identity and lifeworld? The investigators will conduct individual semi-structured qualitative interviews with all the physiotherapists from the IPR interviews.

Criteria for success:

* At least 80% of the patients complete the intervention and the questionnaires after 8-weeks
* At least 80% of the patients' complete questionnaires at 6-month follow-up
* At least 90% of physiotherapists complete the study period
* No adverse events by using the PDB-app
* Patient satisfaction score measured with CSQ-8 ≥20 (indicate good satisfaction)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Obstructive Pulmonary Disease
* Mucus-related issues ≥3 times per week
* Speak and write Norwegian
* Ability to independently operate a smartphone and/or iPad

Exclusion Criteria:

* Severe mental illness
* Substance abuse that hinder participation in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Recruitment rate (n, %)
Intervention adherence | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Intervention adherence (n, %)
Adverse events | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Adverse events (n, %)
Dropout rate | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Dropout (n, %)
Health related outcomes | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  - Dyspnea-12 (D-12) scale score (score 0-36) - low score indicates better outcome
Health related outcomes | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Modified Medical Research Council dyspnea scale (mMRC) (score 0-4) - low score indicates better outcome
Health related outcomes | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Chalder Fatigue Scale (CFQ-11) (score 0-33) - low score indicates better outcome
Health related outcomes | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  COPD Assessment Test (CAT) (score 0-40) - low score indicates better outcome
Health related outcome | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Generalized Anxiety Disorder Assessment (GAD-7) (score 0-21) - low score indicates better outcome
Health related outcome | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Patient Health Questionnaire-9 (PHQ-9) (score 0-27) - low score indicates better outcome
Health related outcomes | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Patient Health Questionnaire-9 (PHQ-9) (score 0-27) - low score indicates better outcome
Health related outcomes | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  EuroQol Questionnaire (EQ-5D) (index and VAS score 0-100) Index: An overall score is generated, ranging from <0 to 1. Low score indicates worse outcome VAS score: low score indicates worse outcome
Physical functioning | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  60 seconds Sit-To-Stand (60sSTS) (number of repetitions) - Higher number of repetitions indicates better outcome
Exacerbations, hospital admissions and use of healthcare services | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  The number of exacerbations, hospital admissions and use of healthcare services (n)
Health literacy | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Health Literacy Questionnaire (HLQ) (44 items, 9 domains) - Health literacy was measured using three domains of the HLQ; 3) Actively managing my health, 6) Ability to engage actively with health-care providers and 9) Understand health information well enough to know what to do. Domains 1-5 are scored 1-4, and domains 6-9 are scored 1-5. Lower score indicates lower levels of health literacy.
Health literacy | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  E-Health Literacy Questionnaire (e-HLQ) (35 items, 7 domains) - E-Health literachy was measured using two domains of the e-HLQ; 3) Ability to actively engage with digital services and 5) Motivated to engage with digital services. Scores range from 1-4. Lower score indicates lower levels of e-Health literacy.
Health education and self-management | From enrollment to end of the treatment at 8 weeks and the end of treatment at 6-month follow-up
  Health Education Impact Questionnaire (heiQ) (48 items, 8 domains) - is used to measure helath edcuation and self-management. We are using three domains of the heiQ; 2) Health related behaviour, 3) Skill and technique acquisition and 5) Self-monitoring and insight. Scores ranges from 1-4. Lower score indicates lower levels of health education impact and self-management.
Satisfaction with treatment | End of treatment at 8 weeks and the end of treatment at 6-month follow-up
  Patients Global Impression of Change (PGIC) (score 0-7) - low score indicates better outcome
Satisfaction with treatment | End of treatment at 8 weeks and the end of treatment at 6-month follow-up
  Client Satisfaction Questionnaire (CSQ-8) (score 8-32) - low score indicates worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bente Frisk, PHD, Principal Investigator — Western Norway University of Applied Sciences
Locations (1):
- Western Norway University of Applied Sciences, Bergen, Norway, Norway

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the approvals granted for this study by the Regional Committee on Medical Research Ethics and the Norwegian Data Inspectorate, the data files will be stored securely and in accordance with the Norwegian Law of Privacy Protection. A subset of the data file with anonymized data will be made available to interested researchers upon reasonable request to Bente Frisk: bente.frisk@hvl.no, providing that Norwegian privacy legislation and the General Data Protection Regulation are respected, and that permission is granted from the Norwegian Data Inspectorate and the data protection officer at Western Norway University of Applied Sciences.
Time Frame: Will be available after data completion of the study: 31.12.30
Access Criteria: In accordance with the approvals granted for this study by the Regional Committee on Medical Research Ethics and the Norwegian Data Inspectorate, the data files will be stored securely and in accordance with the Norwegian Law of Privacy Protection. A subset of the data file with anonymized data will be made available to interested researchers upon reasonable request to Bente Frisk: bente.frisk@hvl.no, providing that Norwegian privacy legislation and the General Data Protection Regulation are respected, and that permission is granted from the Norwegian Data Inspectorate and the data protection officer at Western Norway University of Applied Sciences.